

Title: A Single Center, Open-Label, Phase 1 Study to Evaluate the Pharmacokinetics, Safety and Tolerability of TAK-123 after Intravenous Infusion in Japanese Healthy Adult Male Subjects

NCT Number: NCT04155567

Statistical analysis plan Approve Date: 12-DEC-2019

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).



STUDY NUMBER: TAK-123-1001

A Single Center, Open-Label, Phase 1 Study to Evaluate the Pharmacokinetics, Safety and Tolerability of TAK-123 after Intravenous Infusion in Japanese Healthy Adult Male Subjects

Version: 1st

Date: ^ y to Evaluate the Phanous Infusion in Japane.
Subjects

Version: 1st
Date: 20 December 2019

y:

Prepared by:

Based on:

Protocol Version: Amendment 1 Version

Prote Prote Prote Prote Property of Takeda. Protocol Date: 10 October 2019

Properly of Takeda. For non-confine cial use only and subject to the applicable Tames of use

### TABLE OF CONTENTS 2.0

| 2.0 | TABL | DE OF CONTENTS Oproval Signatures | |
|---|---|---|---|
| 1.1 | Ap | pproval Signatures | .2 |
| 2.0 | TABL | E OF CONTENTS | .3 |
| Lis | st of In- | Text Tables | .4 |
| 3.0 | LIST ( | OF ABBREVIATIONS | .50 |
| 4.0 | OBJE | CTIVES | 26 |
| 4.1 | Pri | mary Objectives | .6 |
| 4.2 | . See | condary Objectives | .6 |
| 4.3 | Stu | imary Objectives | .6 |
| 5.0 | ANAL | Primary Endpoint Secondary Endpoints Safety Endpoints Exploratory Endpoints RMINATION OF SAMPLE SIZE | .7 |
| | 5.1.1 | Primary Endpoint | .7 |
| | 5.1.2 | Secondary Endpoints | .7 |
| | 5.1.3 | Safety Endpoints | .7 |
| | 5.1.4 | Exploratory Endpoints | .7 |
| 6.0 | DETE | RMINATION OF SAMPLE SIZE | .8 |
| 7.0 | MFTF | IODS OF ANALYSIS AND PRESENTATION | () |
| 7.1 | Ge | eneral Principles | .9 |
| | 7.1.1 | Study Definitions | .9 |
| 7.2 | . An | Study Definitions | .9 |
| 7.3 | Dis | sposition of Subjects | 10 |
| | 7.3.1 | Study Information | 10 |
| | 7.3.2 | Screen Failures | 10 |
| | 7.3.3 | Subject Eligibility | 10 |
| | 7.3.4 | Disposition of Subjects | 11 |
| | 7.3.5 | Protocol Deviations and Analysis Sets | |
| 7.4 | De | emographic and Other Baseline Characteristics | 13 |
| 7.5 | X | ldy Drug Exposure and Compliance | |
| 7.6 | Eff | ficacy Analysis | |
| S.1 | 7.6.1 | Primary Efficacy Endpoint(s) | |
| X Olt | 7.6.2 | Secondary Efficacy Endpoint(s) | 14 |
| | 7.6.3 | Additional Efficacy Endpoint(s) | 14 |
| , | 7.6.4 | Statistical/Analytical Issues | 14 |
| 7.7 | Ph | armacokinetic/Pharmacodynamic Analysis | 15 |
| | 7.7.1 | Pharmacokinetic Analysis | |
| | 7.7.2 | Pharmacodynamic Analysis | |
| 7.8 | Sa | fety Analysis | |
| | 7.8.1 | Adverse Events | 17 |
| | 7.8.2 | Clinical Laboratory Evaluations | 20 |

### 3.0 LIST OF ABBREVIATIONS

AΕ adverse event

amount of drug excreted in urine Ae

**ALP** alkaline phosphatase **ALT** alanine aminotransferase **AST** aspartate aminotransferase

aPTT activated partial thromboplastin time **AUC** area under the concentration-time curve

BMI body mass index CL R renal clearance

maximum observed concentration Cmax

**ECG** electrocardiogram

to the applicable reims of Use applicable reims of Use fraction of administered dose of drug excreted in urine fe

gamma glutamyl transferase **GGT** terminal elimination rate constant Lambda z

Medical Dictionary for Regulatory Activities MedDRA

NaBZ sodium benzoate NaPA sodium phenylacetate PK pharmacokinetics prothrombin time PT corrected QT OTc red blood cell **RBC** 

SAE serious adverse event standard deviation SD System Organ Class SOC

**TEAE** treatment-emergent adverse event time of first occurrence of Cmax tmax

t1/2zhalf-life period

WBC WHO Drug volume of distribution during the terminal elimination phase

white blood cell

World Health Organization Drug Dictionary

### 4.0 OBJECTIVES

## 4.1 Primary Objectives

• The primary objective of the study is to evaluate the PK of phenylacetate and benzoate after intravenous infusion of TAK-123 in Japanese healthy adult male subjects.

## 4.2 Secondary Objectives

• The secondary objective of the study is to evaluate the safety and tolerability of TAK-123 after intravenous infusion of TAK-123 in Japanese healthy adult male subjects.

### 4.3 Study Design

This study is a single-center, open-label, uncontrolled study.

In this study, TAK-123 will be administered intravenously as a loading dose over 90 minutes at the dose level of 3.75 g/m<sup>2</sup> of NaPA and 3.75 g/m<sup>2</sup> of NaBZ under the breakfast fasting condition, followed by an equivalent maintenance dose over 24 hours to evaluate the PK, safety and tolerability of TAK-123 in Japanese healthy adult male subjects.

A 4 mg of dose of ondansetron will be administered intravenously 30-40 minutes before the start of TAK-123 infusion.

The dose of TAK-123 to be investigated is shown in Table 4.a. The dose of ondansetron to be administered before the administration of TAK-123 is shown in Table 4.b.

Table 4.a Dosage of TAK-123

| Study drug | Dose | Mode of administration |
|---|---|---|
| TAK-123 | 3.75 g/m <sup>2</sup> of Nal | PA and (1) Intravenous infusion (via a peripheral vein) over 90 minutes as a |
| | $3.75 \text{ g/m}^2 \text{ of Nal}$ | BZ loading dose |
| | Ċ | 2) An equivalent intravenous infusion (via a peripheral vein) over 24 hours as a maintenance dose after the completion of the above 1). |
| | | nous us a manifemente dose after the completion of the doctor). |

Table 4.b Dosage of ondansetron

| Premedication Dose | Mode of administration |
|--------------------|---------------------------|
| Ondansetron 4 mg | Slow intravenous infusion |
| of Takeou | |
| 6 tober | |

### 5.0 ANALYSIS ENDPOINTS

## 5.1.1 Primary Endpoint

G applicable reims of Use the applicable reims of Use • PK parameters (C<sub>max</sub>, AUC<sub>last</sub>, AUC<sub>∞</sub>) of phenylacetate, benzoate, and these metabolites (phenylacetylglutamine and hippurate).

### 5.1.2 Secondary Endpoints

Number of subjects with treatment-emergent adverse events (TEAEs)

## 5.1.3 Safety Endpoints

TEAEs, laboratory tests, vital signs, body weight, and 12-lead ECG

## 5.1.4 Exploratory Endpoints

- Plasma PK parameters  $(t_{max}, t_{1/2z}, \lambda_z)$  of phenylacetate, benzoate, and these metabolites (phenylacetylglutamine and hippurate)
- Property of Takeda. For non-commercial use only and Urinary excretion amounts (Ae) and excretion ratios (fe) of phenylacetate, benzoate, and these metabolites (phenylacetylglutamine and hippurate)

Properly of Takeda, For non-commercial use only and subject to the applicable of the property of takeda.

### **7.0** METHODS OF ANALYSIS AND PRESENTATION

### 7.1 **General Principles**

### 7.1.1 Study Definitions

The following definitions and calculation formulas will be used.

- Treatment-emergent adverse event (TEAE): An adverse event whose date of onset occurs on or after the start of study drug (TAK-123)
- Pretreatment event (PTE): Any untoward medical occurrence in a clinical investigation subject who has signed informed consent to participate in a study but prior to administration of study drug (TAK-123)
- Descriptive statistics: Number of subjects, mean, standard deviation, maximum, minimum, and quartiles
- Coefficient of variation (CV) (%): Standard deviation / mean \* 100

### 7.2 **Analysis Sets**

- nd subi Safety analysis set: All subjects who received at least one dose of TAK-123
- Pharmacokinetic analysis set: All subjects who received at least one dose of TAK-123 Property of Takeda. For non-commercial and provided sufficient PK measurements available to estimate PK parameters, at least 1

### 7.3 **Disposition of Subjects**

### 7.3.1 **Study Information**

All Subjects Who Signed the Informed Consent Form Analysis Set:

**Analysis** 

Variable(s): Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit/Contact

MedDRA Version

SAS Version Used for Creating the Datasets

Analytical

Method(s): (1) Study Information

the applicable terms of Use ion Study information shown in the analysis variables section will be provided.

7.3.2 **Screen Failures** 

All Subjects Who Did Not Receive Study Drug (TAK-123) Analysis Set:

**Analysis** 

Variable(s): Age (years)

Analytical

(1) Screen Failures Method(s):

Descriptive statistics will be provided.

**Subject Eligibility** 

All Subjects Who Signed the Informed Consent Form Analysis Set:

**Analysis** 

Variable(s) Study Drug (TAK-123) [Treated, Not Treated]

**Administration Status** 

Primary Reason for Subject Not [Adverse Event, Death, Lost to

Being Treated Follow-up, Protocol Deviation,

> Sample Size Sufficient, Screen Failure, Study Terminated by Sponsor, Withdrawal by Subject,

Other]

Proberty of Lakeg Analytical

> Method(s): (1) Study Drug (TAK-123) Administration Status

cable Terms of Use Frequency distributions will be provided. When calculating percentages for the primary reasons for subject not being treated, the total number of not treated subjects will be used as the denominator.

### 7.3.4 **Disposition of Subjects**

All Subjects Who Received Study Drug (TAK-123) Analysis Set:

**Analysis** 

[Completed All Planned Study Variable(s): **Study Completion Status** 

Visits, Did Not Complete All

Planned Study Visits]

Reason for Discontinuation of

Follow-up, Protocol Deviation, Study Visits

Sample Size Sufficient, Study

[Adverse Event, Death, Lost to

Terminated by Sponsor, Withdrawal

by Subject, Other]

Analytical

(1) Disposition of Subjects Method(s):

> Frequency distributions will be provided. When calculating percentages for the reasons for discontinuation, the total number of subjects who did not complete all planned study visits will be used as the denominator.

# **Protocol Deviations and Analysis Sets**

### 7.3.5.1 Protocol Deviations

Analysis Set. All Subjects Who Received Study Drug (TAK-123)

Analysis

Variable(s): Significant Protocol [Entry Criteria, Concomitant Medication, Procedure

> Deviation Not Performed Per Protocol, Study Medication,

> > Withdrawal Criteria, Major GCP Violations]

Analytical

Method(s): (1) Protocol Deviations

> Frequency distribution will be provided for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same category will be counted only once.

Properly of Takeda, For non-confiner cial use only and subject to the applicable Terms of Use

## 7.3.5.2 Analysis Sets

All Subjects Who Received Study Drug (TAK-123) Analysis Set:

Analysis

Variable(s): Handling of Subjects

List]

**Analysis Sets** 

Safety Analysis Set [Included] [Included] Pharmacokinetic Analysis Set

Analytical

Method(s): (1) Subjects Excluded from Analysis Sets

(2) Analysis Sets

Frequency distributions will be provided. For (1), a subject who has several reasons for exclusion will be counted once in each appropriate category. A subject who has several reasons for exclusion that can be classified into the same category will be counted only once.

### **Demographic and Other Baseline Characteristics** 7.4

Safety Analysis Set Analysis Set:

**Analysis** 

Variable(s): Age (years)

> Height (cm) Weight (kg)  $BMI (kg/m^2)$

Smoking Classification [Never, Current, Former]

Alcohol Classification [Daily, A Few Times Per Week, A

Few Times Per Month, No]

Caffeine Classification [Yes, No]

(1) Summary of Demographics and Baseline Characteristics

Frequency distributions for categorical variables and descriptive statistics

for continuous variables will be provided.

# 7.6.4.4 Multiple Comparison/Multiplicity

Not applicable

## Use of an "Efficacy Subset" of Subjects

Not applicable.

## 7.6.4.6 Active-Control Studies Intended to Show Equivalence or Non-Inferiority

Not applicable.

### 7.6.4.7 Examination of Subgroups

Not applicable.

## 7.7 Pharmacokinetic/Pharmacodynamic Analysis

### 7.7.1 Pharmacokinetic Analysis

## 7.7.1.1 Plasma Concentrations

Analysis Set: Pharmacokinetic Analysis Set

Analysis

Variable(s): Plasma Concentrations of Phenylacetate, Benzoate and These Metabolites

(Phenylacetylglutamine and Hippurate)

Visit: Predose; 0.25, 0.75, 1.5, 2.5, 4.5, 6.5, 8.5, 10.5, 12.5, 16.5, 25.5, 26, 26.5,

27, 27.5, 28, 28.5, 29.5, 30.5, 32.5 and 48 Hours Postdose;

Analytical

Property of Lakeda. For

Method(s): The following summaries will be provided.

Summary of Plasma Concentrations by Visit
 Descriptive statistics and CV will be provided by visit.

(2) Case Plot of Plasma Concentrations
Plots over time for each subject will be presented. The vertical axis will be a normal scale and a common logarithmic scale.

(3) Mean and Standard Deviation Plot of Plasma Concentrations
Mean and standard deviation will be plotted for each analysis variable.
Visit will be plotted on the horizontal axis and each of the analysis variables will be plotted on the vertical axis. The vertical axis will be a normal scale.

(4) Mean Plot of Plasma Concentrations

Mean will be plotted for each analysis variable. Visit will be plotted on the horizontal axis and each of the analysis variables will be plotted on the vertical axis. The vertical axis will be a common logarithmic scale.

### 7.7.1.2 Pharmacokinetic Parameters

Analysis Set: Pharmacokinetic Analysis Set

Analysis

Variable(s): Pharmacokinetic Parameters of Phenylacetate, Benzoate and These

Metabolites (Phenylacetylglutamine and Hippurate)

AUClast AUCinf AUC48
Cmax tmax t1/2z

Lambda z Vz (for Phenylacetate CL (for Phenylacetate

and Benzoate) and Benzoate)

Analytical

Method(s): The following summary will be provided.

(1) Summary of Pharmacokinetic Parameters
For AUClast, AUCinf, AUC48 and Cmax, descriptive statistics,
geometric mean, CV and geometric CV will be provided. For tmax,
descriptive statistics will be provided. For all other variables,
descriptive statistics and CV will be provided.

## 7.7.1.3 Urine Pharmacokinetic Parameter

Analysis Set: Pharmacokinetic Analysis Set

Analysis

Variable(s): Urine Pharmacokinetic Parameters of Phenylacetate, Benzoate and These

Metabolites (Phenylacetylglutamine and Hippurate)

Urine Pharmacokinetic Parameters of Sum of Phenylacetate and

Phenylacetylglutamine, and Sum of Benzoate and Hippurate for fe48

Ae48 fe48 CLR

Analytical

Method(s): The following summary will be provided.

(1) Summary of Urine Pharmacokinetic Parameter Descriptive statistics and CV will be provided.

### 7.7.2 Pharmacodynamic Analysis

Not applicable.

### 7.8 **Safety Analysis**

In this study, safety will be evaluated as the primary endpoint.

### 7.8.1 Adverse Events

7.8.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

**Analysis** 

Variable(s): **TEAE** 

Relationship to Study Drug (TAK-Categories:

123)

[Related, Not Related] Mild, Moderation Intensity

Analytical

The following summaries will be provided. Method(s):

(1) Overview of Treatment-Emergent Adverse Events

- 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 2) Relationship of Treatment-Emergent Adverse Events to study drug (TAK-123) (number of events, number and percentage of subjects)
- 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 4) Treatment-Emergent Adverse Events leading to study drug (TAK-123) discontinuation (number of events, number and percentage of (subjects)
- Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- Property of Takedai. For non's 6) Relationship of serious Treatment-Emergent Adverse Events to study drug (TAK-123) (number of events, number and percentage of subjects)
  - 7) Serious Treatment-Emergent Adverse Events leading to study drug (TAK-123) discontinuation (number of events, number and percentage of subjects)
  - 8) Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects)

TEAEs will be counted according to the rules below. Percentages will be based on the number of subjects in the safety analysis set.

Number of subjects

- Summaries for 2) and 6)
- A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.

  Summaries other than 2), 3), and 6)

  A subject with multiple of the Teau once in the Related category. • Summary for 3)
- Summaries other than 2), 3), and 6)

## Number of events

For each summary, the total number of events will be calculated.

# 7.8.1.2 Displays of Treatment-Emergent Adverse events

Analysis Set: Safety Analysis Set

Analysis

Variable(s): **TEAE** 

[Mild, Moderate, Severe] Categories: Intensity

Jese Only and subject to Period [Loading Period, Maintenance

Period, After Infusion Period]

Analytical

Probeith of Lakeda.

The following summaries will be provided using frequency distribution. Method(s):

> TEAEs will be coded using the MedDRA and will be summarized using SOC and PT.

SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted Oin decreasing frequency for tables provided by System Organ Class only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (5) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

insofuse

- (6) Intensity of Drug-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
- (7) Treatment-Emergent Adverse Events Leading to Study Drug (TAK-123) Discontinuation by System Organ Class and Preferred Term
- (8) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (9) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term by Period

The frequency distribution will be provided according to the rules below. Percentages will be based on the number of subjects who were treated in the safety analysis set.

## Number of subjects

- Summary tables other than (5) and (6)
  A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT.
- Summary tables for (5) and (6)
  A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity.

# 7.8.1.3 Displays of Pretreatment Events

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis

Variable(s): PTE

Analytical

Method(s): The following summaries will be provided using frequency distribution.

PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

- (1) Pretreatment Events by System Organ Class and Preferred Term
- (2) Serious Pretreatment Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below. Number of subjects

The applicable Terms of Use emails A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in that PT.

### 7.8.2 **Clinical Laboratory Evaluations**

### 7.8.2.1 Hematology and Serum Chemistry

Analysis Set: Safety Analysis Set

**Analysis** 

Variable(s): Hematology

> Red Blood Cell (RBC) Hemoglobin

White Blood Cell **Platelets** 

(WBC)

WBC Differentials (Neutrophils, Eosinophils, Basophils, Lymphocytes,

Monocytes)

PT

Serum Chemistry

Albumin **Total Protein** Blood Urea Nitrogen

Total Bilirubin Creatinine Direct Bilirubin

Sodium Potassium Chloride

ALP Calcium Creatine kinase

**AST ALT GGT** 

Glucose Glucose

(Self-monitoring)

Glucose (Self-monitoring): Visit:

Predose; 1 and 1.5 Hours Postdose;

Sodium, Potassium and Chloride:

Predose; 1.5, 25.5, and 48 Hours Postdose; Day 8

Variables other than Glucose (Self-monitoring), Sodium, Potassium and

Chloride:

Predose; 25.5, and 48 Hours Postdose; Day 8

(Data obtained at Day -1 will be used as the "Predose" visit)

Property of Takeda The following summaries will be provided.

(1) Summary of Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline (each postdose visit - Predose) will be provided by visit.

- (2) Case Plots of Laboratory Test Results Plots over time for each subject will be presented.
- reims of Use (3) Summary of Shifts of Laboratory Test Results Shift tables showing the number of subjects in each category at Predose and each postdose visit will be provided.

For each laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range. The shift tables will be based on these classifications.

# 7.8.2.2 Urinalysis

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Specific Gravity

рΗ

Protein Glucose

Occult blood **Nitrite** 

Urobilinogen

Predose; 25.5, and 48 Hours Postdose; Day 8 Visit:

(Data obtained at Day -1 will be used as the "Predose" visit)

Analytical

For specific gravity, summaries (1), (2) and (4) will be provided. Property of Takeda Method(s):

For each variable other than specific gravity, summaries (3) and (4) will be provided.

- (1) Summary of Urine Laboratory Test Results and Change from Baseline by Visit
  - Descriptive statistics for observed values and changes from baseline (each postdose visit - Predose) will be provided by visit.
- (2) Case Plots of Urine Laboratory Test Results Plots over time for each subject will be presented.

- (3) Number of Subjects in Categories of Urine Laboratory Test Results
- Shift tables showing the number of subjects in each category at Predose and each postdose visit will be provided. The laboratory value for specific gravity will be classified as "Low" "Extraction of the companies of the compani (4) Summary of Shifts of Urine Laboratory Test Results value for each urine laboratory test other than specific gravity will be classified as "Normal" or "Abnormal" relative to the normal reference range. The shift tables will be based on these classifications. and subject

### 7.8.2.3 Blood Gas Test

Analysis Set: Safety Analysis Set

Analysis

Variable(s): pН

Predose; 1.5 and 25.5 Hours Postdose; Visit:

(Data obtained at Day -1 will be used as the "Predose" visit)

Analytical

The following summaries will be provided. Method(s):

> (1) Summary of Blood Gas Test Results and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline (each postdose visit - Predose) will be provided by visit.

(2) Case Plots of Laboratory Test Results Plots over time for each subject will be presented.

# Vital Signs and Weight

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Temperature

> Systolic Blood Pressure Diastolic Blood Pressure

Respiration Rate

Pulse Rate

Visit:

Analytical

Method(s):

The following summaries will be provided.

(1) Summary of Vital Signs Parameters and Weight and Change from Baseline by Visit

Descriptive statistics for observed values and change (each postdose visit - Predose) will be -
2) Case Plots of Vital Signs P

Plots over time

ercial use only and sur

### 7.8.4 12-Lead ECGs

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Heart Rate

RR Interval

PR Interval

QRS Interval

QT Interval

**QTcF** Interval

Interpretation [Within Normal Limits, Abnormal but not

Clinically Significant, Abnormal and

Clinically Significant]

Predose, 1.5 and 48 Hours Postdose; Day 8

Analytical Method(s): For each variable other than 12-lead ECG interpretations, summaries (1)

and (2) will be provided.

For 12-lead ECG interpretation, summary (3) will be provided.

(1) Summary of ECG Parameters and Change from Baseline by Visit Descriptive statistics for observed values and changes from baseline (each postdose visit - Predose) will be provided by visit.

- (2) Case Plots of ECG Parameters Plots over time for each subject will be presented.
- the ar (3) Summary of Shift of 12-lead ECG Interpretation Shift table showing the number of subjects in each category at "Predose" visit and each postdose visit will be provided.

## 7.8.5 Other Observations Related to Safety

Not applicable.

### 7.9 **Interim Analysis**

Not applicable.

## **Changes in the Statistical Analysis Plan**

differ from and see only and se The analyses in the statistical analysis plan do not differ from the analyses specified in the

Properly of Takeda, For non-confine cial use only and subject to the applicable Taines of Use